CLINICAL TRIAL: NCT03301532
Title: Compatibility of Triheptanoin (C7) With the Ketogenic Diet in Patients Diagnosed With Glucose Transporter Type 1 Deficiency
Brief Title: Compatibility of C7 With Ketogenic Diet in Patients Diagnosed With G1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Juan Pascual, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102015-091; R01NS094257-01A1 (NIH)
Record Dates: First submitted 2017-08-29; First posted 2017-10-04 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: GLUT1DS1
Keywords: G1D, glucose, transporter
MeSH Terms: interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients on a ketogenic diet (Experimental): This is a one arm study were patients will be receiving an oil called triheptanoin. Patients will be consuming triheptanoin 4 times over the course of one day. The triheptanoin oil will take up 45% of their daily calories on the day the day they are taking the oil.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Dietary supplementation with triheptanoin
  Other Names: C7 oil

SUMMARY:
To explore triheptanoin (C7 oil) compatibility with the ketogenic diet by evaluating EEG, and seizure rate, glycemia and ketosis in proven G1D patients receiving a ketogenic diet.

DETAILED DESCRIPTION:
This is a single site, open label proof of principle exploratory trial to investigate the compatibility of C7 oil with the ketogenic diet in subjects diagnosed with G1D. The ketogenic diet will have been previously described by the patient's treating physician independently of this study and for clinical reasons. The ketogenic diet supplies over 50% of calories from fat, subjects, who are already tolerating over this much fat as part of their previously prescribed ketogenic diet, will replace 45% of their daily caloric intake with the triheptanoin for 24 hours, during a 48 hour inpatient stay. Subjects will have a continuous EEG to monitor for any potential C7 related changes in seizure before, during, and after triheptanoin oil ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glucose transporter type 1 deficiency (G1D), confirmed by clinical genotyping at a CLIA-certified laboratory.
* Stable on ketogenic diet at 2.5:1 to 4:1 ratio (i.e., no changes in ratio will have taken place for 2 months). The initiation of a ketogenic diet is previous to - and thus is not part of this study.
* Males and females 30 months to 35 years and 11 months old inclusive.

Exclusion Criteria:

* Subjects with evidence of independent, unrelated metabolic and/or genetic disease.
* Subjects with a chronic gastrointestinal disorder, such as irritable bowel syndrome, crohn's disease, or colitis that could increase the subject's risk of developing diarrhea or stomach pain.
* Subjects with a BMI (body mass index) greater than or equal to 30.
* Subjects currently not on ketogenic diet.
* Women who are pregnant or breast feeding may not participate. Women who plan to become pregnant during the course of the study, or who are unwilling to use birth control to prevent pregnancy (including abstinence) may not participate. Females age 10 and over will be asked to provide a urine sample for a pregnancy test via dipstick. Subjects will be asked to agree to abstinence or another form of birth control for the duration of the study.
* Allergy/sensitivity to C7
* Previous use of triheptanoin less than 1 month prior to study initiation.
* Treatment with medium chain triglycerides in the last 24 hours.
* Subjects exhibiting signs of dementia, or diagnosed with any degenerative brain disorder (such as Alzheimer's disease) that would confound assessment of cognitive changes, in the opinion of the investigator.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent, or assent for children age 10-17,
* Addition of a new antiseizure drug in the previous 3 months.

Ages: 30 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pascual, M.D., Principal Investigator — Study Principal Investigator
Locations (1):
- UTexasSouthwestern, Dallas, Texas, United States

REFERENCES:
- [Result] Avila A, Malaga I, Sirsi D, Kayani S, Primeaux S, Kathote GA, Jakkamsetti V, Kallem RR, Putnam WC, Park JY, Shinnar S, Pascual JM. Combination of triheptanoin with the ketogenic diet in Glucose transporter type 1 deficiency (G1D). Sci Rep. 2023 Jun 2;13(1):8951. doi: 10.1038/s41598-023-36001-x. PMID 37268656

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Triheptanoin (C7): Triheptanoin (C7 oil, liquid). Subjects consumed triheptanoin 4 times over the course of one day. The approach included substituting a fraction of ketogenic diet fat with C7, weight by weight, at the maximum tolerable dose (45% of their their daily calories) in individuals receiving a ketogenic diet prior to enrolment prescribed independently of this study.
Period: Overall Study
Arm/Group | Experimental: Triheptanoin (C7)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Triheptanoin (C7 Oil, Liquid): C7 oil was given at maximum tolerated dose (45% of total daily calories) to 10 Glut1 subjects receiving a ketogenic diet prior to enrolment as medically prescribed independently of this study.
Arm/Group | Triheptanoin (C7 Oil, Liquid)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
  Argentina | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Ketosis (Beta-hydroxybutyrate Levels)
Description: Change in Ketosis as measured by changes in blood beta-hydroxybutyric acid levels.
Time Frame: Day 1, Day 4
Population: Subjects with Glut1 deficency
Measure: Mean (Standard Deviation); unit: mM
Groups:
- Ketosis: Participants BHB levels were checked daily on days 1 - 4. Treatment: Triheptanoin (C7), orally, dose of 45% of the total daily calories divided in four equally spaced administrations (i.e., one dose every 4 hours to a total of four doses in one day).
Arm/Group | Ketosis
Number analyzed (Participants) | 10
mM | 3.82 (1.9)

2. Secondary Outcome: Fraction of Subjects (of a Total of 10 Studied) Who Exhibit a Change in Observable Seizure Rate
Description: The percent change in observable seizure rate is measured as the change in observable seizure numbers from baseline to Day 4.
  Seizure rate is defined as count of seizures per patient per day.
Time Frame: Baseline (Day 1) - Day 4
Population: All subjects with Glut1 deficiency studied. Triheptanoin (C7 oil, liquid). Subjects consumed triheptanoin 4 times over the course of one day. The approach included substituting a fraction of ketogenic diet fat with C7, weight by weight, at the maximum tolerable dose (45% of their their daily calories) in individuals receiving a ketogenic diet prior to enrolment prescribed independently of this study.
Measure: Count of Participants; unit: Participants
Groups:
- Fraction of Subjects With a Change in Seizure Rate: Ratio of subjects with seizure rate changes divided by total number of subjects. The seizure rate is based on changes in observable seizure numbers.
Arm/Group | Fraction of Subjects With a Change in Seizure Rate
Number analyzed (Participants) | 10
Participants | 3

3. Secondary Outcome: Change in Glycemia
Description: Change in Glycemia is measured as changes in blood glucose levels.
Time Frame: Day 1 - Day 4
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Glycemia: Changes in blood glucose levels.
Arm/Group | Glycemia
Number analyzed (Participants) | 10
mg/dl | 81.2 (13.6)

ADVERSE EVENTS:
Time Frame: Days 1 - 4
Groups:
- Ketosis: Participants BHB levels were checked daily on days 1 - 4.
Arm/Group | Ketosis
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketosis (N=10)
Seizures (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03301532/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03301532/ICF_001.pdf